CLINICAL TRIAL: NCT01572545
Title: Comparative Effect of Zoledronic Acid Versus Denosumab on Serum Sclerostin Levels of Postmenopausal Women With Low Bone Mass: A Multicenter, Randomized, Head-to-head Clinical Trial
Brief Title: Comparative Effect of Zoledronic Acid Versus Denosumab on Serum Sclerostin of Postmenopausal Women With Low Bone Mass
Acronym: DenoZol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: 424 General Military Hospital (Other); 251 Hellenic Air Force & VA General Hospital (Other)
Responsible Party: Principal Investigator, Stergios A. Polyzos, MD, MSc, PhD, Principal Investigator, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PolyzosAnastasilakis
Record Dates: First submitted 2012-04-03; First posted 2012-04-06 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Postmenopausal Osteoporosis
Keywords: bone turnover; denosumab; postmenopausal osteoporosis; sclerostin; zolendronic acid
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Sclerosteosis | interventions — Denosumab; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Denosumab (Experimental)
  Interventions: Drug: Denosumab
- Zoledronic Acid (Experimental)
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Denosumab — Denosumab (injection), 60 mg, administered as a single subcutaneous injection once
  Other Names: Prolia
  Arms: Denosumab
Drug: Zoledronic acid — Zoledronic acid (vial), 5 mg, administered once as a single 15- to 30-minute intravenous infusion
  Other Names: Aclasta
  Arms: Zoledronic Acid

SUMMARY:
The primary aim of the study is the comparative effect of zolendronic acid versus denosumab on serum sclerostin levels in postmenopausal women with low bone mass.

Secondary aims are their comparative effect on serum dickkopf-1, osteoprotegerin, receptor activator of nuclear factor kappaB ligand (RANKL) and bone turnover markers (procollagen type I N-terminal peptide [PINP] and C-terminal cross-linking telopeptide of type I collagen [CTX]).

DETAILED DESCRIPTION:
Osteoporosis is the most common bone disease, caused by a relatively increased rate of bone resorption by the osteoclasts that exceeds the rate of bone formation by the osteoblasts, resulting in net loss of bone mass. To-date, antiresorptive agents, which inhibit osteoclast activity and induce their apoptosis, are considered as the cornerstone of osteoporosis prevention and treatment.

Bisphosphonates currently represent the first line antiresorptive agents for the management of postmenopausal osteoporosis. Zoledronic acid is considered to-date the most potent bisphosphonate. A once-yearly infusion of intravenous zoledronic acid decreases bone turnover, improves bone density and decreases the vertebral and non-vertebral fracture risk.

Most recently, denosumab (AMG-162) has been launched for the treatment of postmenopausal osteoporosis. Denosumab, a fully human monoclonal IgG2 antibody against human RANKL, specifically binds and neutralizes the receptor activator of nuclear factor kappaB ligand (RANKL) in order to decrease bone resorption and subsequent bone loss. Subcutaneous administration of denosumab every six months decreases bone turnover markers, increases bone mineral density and reduces the vertebral and non-vertebral fracture risk.

The role of sclerostin in bone metabolism is emerging. Sclerostin is the secreted expression of the SOST gene. In adult human bone, sclerostin is expressed only by osteocytes and inhibits bone formation by osteoblasts. It has been proposed that sclerostin expression by newly embedded osteocytes at the onset of osteoid mineralization may serve as a negative feedback signal on osteoblasts to prevent overfilling of the basic multicellular unit.

Although zoledronic acid and denosumab are currently regarded as the most potent antiresorptive agents, there is no head-to-head comparative study. This study primarily aims to the comparative effect of zoledronic acid and denosumab on serum sclerostin levels and secondarily on serum dickkopf-1, osteoprotegerin, RANKL and bone turnover markers (procollagen type I N-terminal peptide [PINP] and C-terminal cross-linking telopeptide of type I collagen [CTX]).

ELIGIBILITY:
Inclusion Criteria:

* Caucasian postmenopausal women older than 40 years
* Low bone mass at lumbar spine (L2-L4) or femoral neck (BMD T-score of ≤ -2.0) or BMD T-score of > -2.0 coexistent with low-energy fracture of vertebral, femoral neck or forearm
* Patient's informed consent to participate

Exclusion Criteria:

* Secondary osteoporosis
* Any bone and mineral disorder other than osteoporosis, including primary or secondary hyperparathyroidism, Paget's disease of bone, osteogenesis imperfecta, rheumatologic diseases, paraplegia, chronic immobilization
* Severe liver or kidney disease (creatinine clearance < 60ml/min/1.73m2) or liver or kidney transplantation
* Premature ovarian failure
* Uncontrolled thyroid disease
* Any malignancy
* Any musculoskeletal injury or surgical procedure 6 months prior to baseline
* Dental surgery or teeth removed 3 months prior to baseline or plan to
* History or concomitant medications that could affect bone metabolism, including immunosuppressive, anticonvulsant, antiviral and anti-tuberculosis agents, addictive drugs, corticosteroids, non-steroidal anti-inflammatory drugs, amiodarone, thiazolidinediones, interferon, metronidazole, and tamoxifen

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Sclerostin | 12 weeks
  Serum sclerostin levels

SECONDARY OUTCOMES:
Dickkopf-1 | 12 weeks
  Serum dickkopf-1 (DKK-1) levels
OPG/RANKL | 12 weeks
  Serum osteoprotegerin (OPG) and receptor activator of nuclear factor kappaB ligand (RANKL) levels
Calcium metabolism | 12 weeks
  Serum calcium, phosphate, intact parathyroid hormone (PTH) and 25-hydroxy-vitamin D (25OHD)
Bone turnover | 12 weeks
  Serum bone turnover markers (total alkaline phosphatase [TSAP], type I N-terminal peptides [PINP] και C-terminal cross-linking telopeptide of type I collagen [CTX])

CONTACTS AND LOCATIONS:
Overall Officials: Stergios A Polyzos, MD, MSc, PhD, Principal Investigator — Aristotle University Of Thessaloniki; Athanasios D Anastasilakis, MD, PhD, Principal Investigator — 424 General Military Hospital; Polyzois Makras, MD, PhD, Principal Investigator — 251 Hellenic Air Force & VA General Hospital
Locations (3):
- Greece (3):
  - 251 Hellenic Air Force Hospital, Athens, Attikis
  - 424 General Military Hospital, Thessaloniki, Thessaloniki
  - Second Medical Clinic, Medical School, Aristotle University of Thessaloniki, Ippokration Hospital, Thessaloniki, Thessaloniki

REFERENCES:
- [Background] Anastasilakis AD, Polyzos SA, Makras P, Sakellariou GT, Bisbinas I, Gkiomisi A, Delaroudis S, Gerou S, Ballaouri I, Oikonomou D, Papapoulos SE. Acute phase response following intravenous zoledronate in postmenopausal women with low bone mass. Bone. 2012 May;50(5):1130-4. doi: 10.1016/j.bone.2012.02.006. Epub 2012 Feb 15. PMID 22366634
- [Background] Anastasilakis AD, Polyzos SA, Anastasilakis CD, Toulis KA, Makras P. Denosumab and bisphosphonates: rivals or potential "partners"? A "hybrid" molecule hypothesis. Med Hypotheses. 2011 Jul;77(1):109-11. doi: 10.1016/j.mehy.2011.03.039. Epub 2011 Apr 8. PMID 21482033
- [Background] Polyzos SA, Anastasilakis AD, Bratengeier C, Woloszczuk W, Papatheodorou A, Terpos E. Serum sclerostin levels positively correlate with lumbar spinal bone mineral density in postmenopausal women--the six-month effect of risedronate and teriparatide. Osteoporos Int. 2012 Mar;23(3):1171-6. doi: 10.1007/s00198-010-1525-6. Epub 2011 Jan 11. PMID 21305266
- [Background] Anastasilakis AD, Toulis KA, Polyzos SA, Terpos E. RANKL inhibition for the management of patients with benign metabolic bone disorders. Expert Opin Investig Drugs. 2009 Aug;18(8):1085-102. doi: 10.1517/13543780903048929. PMID 19558335
- [Background] Anastasilakis AD, Toulis KA, Goulis DG, Polyzos SA, Delaroudis S, Giomisi A, Terpos E. Efficacy and safety of denosumab in postmenopausal women with osteopenia or osteoporosis: a systematic review and a meta-analysis. Horm Metab Res. 2009 Oct;41(10):721-9. doi: 10.1055/s-0029-1224109. Epub 2009 Jun 17. PMID 19536731